CLINICAL TRIAL: NCT00138164
Title: A Phase II Multicenter Study of Ontak® (Denileukin Diftitox) in Patients With Relapsed or Refractory B-Cell Non-Hodgkin's Lymphoma
Brief Title: Denileukin Diftitox in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: LIGAND-PIND-123; UCLA-0412087-01; CDR0000439451 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2008-11

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent small lymphocytic lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — denileukin diftitox

INTERVENTIONS:
Biological: denileukin diftitox

SUMMARY:
RATIONALE: Biological therapies, such as denileukin diftitox, may be able to carry cancer-killing substances directly to non-Hodgkin's lymphoma cells.

PURPOSE: This phase II trial is studying how well denileukin diftitox works in treating patients with relapsed or refractory B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of denileukin diftitox, in terms of objective response and time to progression, in patients with relapsed or refractory B-cell non-Hodgkin's lymphoma.

Secondary

* Determine the safety of this drug in these patients.
* Determine the 1-year overall survival of patients treated with this drug.

OUTLINE: This is an open-label, multicenter study.

Patients receive denileukin diftitox IV over 20-80 minutes on days 1-3, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85, 92, and 99 (weeks 1-16) in the absence of disease progression or unacceptable toxicity. Patients achieving a partial response at week 16 may continue treatment once monthly for up to 8 additional doses or until a complete response (CR) is achieved. Patients achieving a CR (at any time) receive 2 additional monthly doses of denileukin diftitox beyond CR.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 25-50 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed B-cell non-Hodgkin's lymphoma (NHL) of 1 of the following subtypes:

  * Diffuse large B-cell lymphoma
  * Follicular lymphoma (grades 1-3)
  * Small lymphocytic lymphoma
  * Transformed B-cell lymphoma
* Relapsed or refractory disease

  * Disease failed to respond to or progressed after ≥ 2 prior treatment regimens (e.g., high-dose therapy [HDT] with stem cell transplantation [SCT]*) NOTE: *Patients who have received HDT with SCT are considered to have diminished bone marrow reserve
* Diminished bone marrow reserve AND/OR mild to moderate cytopenia, meeting 1 of the following criteria:

  * Absolute neutrophil count ≥ 1,000/mm^3 but < 1,500/mm^3 (growth factor independent)
  * WBC ≥ 2,000/mm^3 but < 4,000/mm^3 (growth factor independent)
  * Platelet count ≥ 40,000/mm^3 (25,000/mm^3 if thrombocytopenia is secondary to marrow involvement by lymphoma) but < 150,000/mm^3 (platelet transfusion independent)
* At least 1 bidimensionally measurable lymph node or tumor mass ≥ 4 cm

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 16 weeks

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2 times ULN
* Albumin ≥ 3.0 g/dL
* No history of veno-occlusive disease of the liver
* No chronic hepatitis

Renal

* Creatinine < 2 times ULN

Cardiovascular

* No congestive heart failure
* No New York Heart Association class III-IV cardiac disease
* No ventricular tachycardia
* No fibrillation
* No myocardial infarction within the past 12 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known HIV positivity
* No active GVHD ≥ grade 2 within the past 6 months
* No other serious medical illness or active infection that would preclude study participation
* No known hypersensitivity to denileukin diftitox or any of its components (e.g., diphtheria toxin, interleukin-2, or their excipients)
* No other malignancy within the past 5 years except successfully treated carcinoma in situ of the cervix or basal cell carcinoma

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* At least 6 months since prior allogeneic SCT
* No concurrent immunotherapy

Chemotherapy

* No concurrent chemotherapy

Endocrine therapy

* No concurrent anticancer hormonal therapy
* No concurrent corticosteroids for the treatment of NHL
* Concurrent corticosteroids allowed for the following conditions:

  * Tapering doses of corticosteroids for resolving graft-versus-host disease (GVHD)
  * Low-dose maintenance corticosteroids for the treatment of an autoimmune disorder
  * Corticosteroids as premedication prior to denileukin diftitox administration or as transient treatment for hypersensitivity reactions

Radiotherapy

* More than 4 weeks since prior and no concurrent radiotherapy
* No prior radiotherapy to the only site of evaluable disease unless disease progression has occurred at that site

Surgery

* Not specified

Other

* At least 3 weeks since prior antilymphoma therapy
* More than 4 weeks since prior and no other concurrent experimental therapy, including approved drugs tested in an investigational setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-12; Primary Completion 2006-02 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Objective clinical response (complete or partial response)

SECONDARY OUTCOMES:
Time to progression
Overall survival at 1 year
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Lauren C. Pinter-Brown, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States